CLINICAL TRIAL: NCT00004604
Title: A Phase I Study of Active Immunotherapy With Carcinoembryonic Antigen RNA-Pulsed, Autologous Human Cultured Dendritic Cells in Patients With Metastatic Malignancies Expressing Carcinoembryonic Antigen
Brief Title: Biological Therapy in Treating Patients With Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Morse, MD, Principal Investigator, Duke University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065619; 1817 (Other: Duke IRB)
Record Dates: First submitted 2000-05-02; First posted 2004-04-28 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer; Colorectal Cancer; Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Gastric Cancer; Head and Neck Cancer; Liver Cancer; Lung Cancer; Metastatic Cancer; Ovarian Cancer; Pancreatic Cancer; Testicular Germ Cell Tumor
Keywords: stage IV colon cancer; stage IV breast cancer; recurrent breast cancer; stage IV gastric cancer; recurrent gastric cancer; recurrent non-small cell lung cancer; recurrent pancreatic cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; inflammatory breast cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; unresectable gallbladder cancer; recurrent gallbladder cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; thyroid gland medullary carcinoma; stage IV non-small cell lung cancer; stage IV salivary gland cancer; recurrent salivary gland cancer; Paget disease of the breast with invasive ductal carcinoma; adult primary hepatocellular carcinoma; testicular yolk sac tumor; lung metastases; liver metastases; cholangiocarcinoma of the gallbladder; cholangiocarcinoma of the extrahepatic bile duct; male breast cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Bile Duct Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Liver Neoplasms; Lung Neoplasms; Neoplasm Metastasis; Ovarian Neoplasms; Pancreatic Neoplasms; Testicular Germ Cell Tumor; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Rectal Neoplasms; Inflammatory Breast Neoplasms; Carcinoma, Ovarian Epithelial; Small Cell Lung Carcinoma; Testicular Neoplasms; Carcinoma, Medullary; Salivary Gland Neoplasms; Carcinoma, Hepatocellular; Endodermal Sinus Tumor; Breast Neoplasms, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CEA RNA-pulsed DC cancer vaccine (Experimental): carcinoembryonic antigen RNA-pulsed dendritic cells
  Interventions: Biological: CEA RNA-pulsed DC cancer vaccine

INTERVENTIONS:
Biological: CEA RNA-pulsed DC cancer vaccine — carcinoembryonic antigen RNA-pulsed dendritic cells

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Phase I trial to study the effectiveness of biological therapy in treating patients who have metastatic cancer that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and dose limiting toxicity of an intravenous vaccine of autologous, cultured, dendritic cells pulsed with carcinoembryonic antigen (CEA) RNA in patients with metastatic adenocarcinoma expressing CEA. II. Assess the cellular immune response to the CEA protein. III. Assess the clinical and biochemical response to the treatment and the duration of such response.

OUTLINE: This a three tiered, open label, uncontrolled, dose escalation study. The first 3 patients receive a low dose of intravenous carcinoembryonic antigen (CEA) RNA-pulsed autologous dendritic cells (DC) at weeks 0, 1, 2, and 3. Patients are evaluated for dose limiting toxicity (DLT), immune response, and the antitumor response for at least 1 week before dose escalation may proceed. If there is no DLT in the first three, the next 3 patients are treated at a medium dose of CEA RNA-pulsed autologous DC at 0, 1, 2, and 3 weeks. Finally, if DLT is not seen at the medium dose, the final 6 patients receive intravenous infusions of a high dose of CEA RNA-pulsed autologous DC at weeks 0, 1, 2, and 3. If 1-2 patient(s) experience DLT at the either the low or medium dose levels, 3 more patients are entered at the same dose. If no further DLT occurs, then dose escalation continues. As soon as 3 toxic events occur in 3-6 patients at one dose level, accrual at that level ceases. The MTD is defined as the dose level immediately below that at which more than 3 of 6 patients develop DLT.

PROJECTED ACCRUAL: A minimum of 3 and a maximum of 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic adenocarcinoma expressing carcinoembryonic antigen (CEA) that has failed conventional therapy Measurable or evaluable disease May include elevated CEA level No previously irradiated or known new CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Greater than 6 months Hematopoietic: WBC at least 3,000/mm3 Absolute lymphocyte count at least 1,000/mm3 Hemoglobin at least 9 g/dL Platelet count at least 100,000/mm3 PT less than 1.25 times normal limit PTT less that 1.66 times normal limit Fibrinogen greater than 0.75 times normal limit Hepatic: Bilirubin less than 2.0 mg/dL Renal: Creatinine less than 2.5 mg/dL Cardiovascular: No NYHA class III or IV Pulmonary: FEV1 greater than 70% of predicted FVC greater than 70% of predicted DLCO greater than 70% of predicted No asthma or chronic obstructive pulmonary disease Other: No active or chronic infection (including urinary tract infection) No viral hepatitis HIV negative No concurrent second malignancy other than nonmelanoma skin cancer or controlled superficial bladder cancer No hepatic disease No history of other autoimmune disease such as inflammatory bowel disease, systemic lupus erythematous, ankylosing spondylitis, scleroderma, or multiple sclerosis

PRIOR CONCURRENT THERAPY: Must have recovered from all acute toxic effects Biologic therapy: No concurrent biologic therapy At least 6 weeks since biologic therapy No concurrent immunotherapy No more than 1 prior biologic regimen Chemotherapy: No concurrent chemotherapy At least 6 weeks since chemotherapy No more than 1 prior chemotherapy regimen Endocrine therapy: At least 6 weeks since steroid therapy Radiotherapy: No concurrent radiotherapy At least 12 weeks since therapy including Sr 89 At least 6 weeks since other radiotherapy No prior cranial radiotherapy Surgery: Not specified Other: No concurrent immunosuppressives such as azathioprine or cyclosporine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 1997-02; Primary Completion 2001-06 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Safety | 12 months
  To determine the safety and dose limiting toxicity of intravenous injections of autologous, cultured, dendritic cells pulsed with CEA RNA.

SECONDARY OUTCOMES:
Immune response | 12 weeks
  Evaluation of cellular immune response to the CEA protein. Evaluation of clinical and biochemical response to the treatment and the duration of such response

CONTACTS AND LOCATIONS:
Overall Officials: Herbert K. Lyerly, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States